CLINICAL TRIAL: NCT02016014
Title: Effectiveness of the Use of a Mobile Tool Added to a Standard Intervention in Improving Lifestyles in Adults
Brief Title: Effectiveness of the Use of a Mobile Tool in Improving Lifestyles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI13/00618; GRS 770/B/13 (Registry Identifier: EVIDENT II)
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2016-08

CONDITIONS: Healthy Subjects Without Cardiovascular Disease
Keywords: Physical activity; Alimentation; Information and communication Technology; Arterial aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Lifestyle counseling in physical activity and alimentation and add for three months a smartphopne with a app (EVIDENT) to improve alimentation and physical activity
  Interventions: Device: Smartphone with APP; Behavioral: Counseling on lifestyles
- Lifestyle counseling (Active Comparator): Lifestyle counseling in physical activity and alimentation
  Interventions: Behavioral: Counseling on lifestyles

INTERVENTIONS:
Device: Smartphone with APP — Smartphone with APP (EVIDENT) for 3 months
  Arms: Intervention group
Behavioral: Counseling on lifestyles — Counseling on physical activity and mediterranean diet

SUMMARY:
Objectives: To develop and validate a mobile tool for use in Smartphone supports as a first step, and to evaluate the effect of adding this new tool of information and communication technologies (ICT), to a standardized intervention to increase adherence to nutritional recommendations of the Mediterranean diet and increase physical activity as primary endpoint. Analyze adherence and intervention results from a gender perspective. Methodology: Multicenter, randomized double-blind, clinical trial with two parallel group, aimed at assessing the effects of adding an TIC tool, developed for the Smartphone application (intervention), in support of behavioral and educational recommendations (control) in the increased physical activity and adaptation to the Mediterranean dietary pattern. Population: 1215 included subjects younger than 70 years from the project EVIDENT who agree to participate. Measurement and interventions: Physical activity will be assessed with the accelerometer and the 7-PAR day and adaptation to the Mediterranean diet with a questionnaire of adherence and a food frequency survey. It will also assess vascular structure and function, central blood pressure, Augmentation index, pulse rate and of carotid intima-media thickness. The counsel to adaptation the Mediterranean diet (based on the project PREDIMED) and exercise (based on PEPAF project), will be common to both groups. The intervention group will be added training and use of an application on a Smartphone designed to promote healthy eating and increased physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects since 20 to 70 years

Exclusion Criteria:

Older than 70 years are excluded, due to difficulties in the use of ICTs and those who can not exercise or follow a diet Mediterranean diet

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mediterranean diet compliance | 1 year
  Measurement by medierranean diet questionary from PREDIMED study

SECONDARY OUTCOMES:
Increase physical activity | 1 year
  Measurement by accelerometer and evaluate bay counts/minute

OTHER OUTCOMES:
Cardio ankle vascular index (CAVI) | 1 year
  Measurement by Vasera device

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia-Ortiz, MD, Principal Investigator — Instituto Biosanitario de Salamanca
Locations (1):
- Instituto Biosanitario de Salamanca. Research unit La Alamedilla, Salamanca, Spain

REFERENCES:
- [Background] Garcia-Ortiz L, Recio-Rodriguez JI, Martin-Cantera C, Cabrejas-Sanchez A, Gomez-Arranz A, Gonzalez-Viejo N, Iturregui-San Nicolas E, Patino-Alonso MC, Gomez-Marcos MA; EVIDENT Group. Physical exercise, fitness and dietary pattern and their relationship with circadian blood pressure pattern, augmentation index and endothelial dysfunction biological markers: EVIDENT study protocol. BMC Public Health. 2010 May 6;10:233. doi: 10.1186/1471-2458-10-233. PMID 20459634
- [Background] Grandes G, Sanchez A, Sanchez-Pinilla RO, Torcal J, Montoya I, Lizarraga K, Serra J; PEPAF Group. Effectiveness of physical activity advice and prescription by physicians in routine primary care: a cluster randomized trial. Arch Intern Med. 2009 Apr 13;169(7):694-701. doi: 10.1001/archinternmed.2009.23. PMID 19364999
- [Result] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Derived] Gonzalez-Sanchez J, Recio-Rodriguez JI, Fernandez-delRio A, Sanchez-Perez A, Magdalena-Belio JF, Gomez-Marcos MA, Garcia-Ortiz L; On behalf the EVIDENT Investigators group. Using a smartphone app in changing cardiovascular risk factors: A randomized controlled trial (EVIDENT II study). Int J Med Inform. 2019 May;125:13-21. doi: 10.1016/j.ijmedinf.2019.02.004. Epub 2019 Feb 12. PMID 30914176
- [Derived] Recio-Rodriguez JI, Rodriguez-Martin C, Gonzalez-Sanchez J, Rodriguez-Sanchez E, Martin-Borras C, Martinez-Vizcaino V, Arietaleanizbeaskoa MS, Magdalena-Gonzalez O, Fernandez-Alonso C, Maderuelo-Fernandez JA, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Investigators. EVIDENT Smartphone App, a New Method for the Dietary Record: Comparison With a Food Frequency Questionnaire. JMIR Mhealth Uhealth. 2019 Feb 8;7(2):e11463. doi: 10.2196/11463. PMID 30735141
- [Derived] Gomez-Marcos MA, Patino-Alonso MC, Recio-Rodriguez JI, Agudo-Conde C, Romaguera-Bosch M, Magdalena-Gonzalez O, Gomez-Arranz A, Mendizabal-Gallastegui N, Angel Fernandez-Diez J, Gomez-Sanchez L, Maderuelo-Fernandez JA, Rodriguez-Sanchez E, Garcia-Ortiz L; on behalf the EVIDENT Investigators 11. Short- and long-term effectiveness of a smartphone application for improving measures of adiposity: A randomised clinical trial - EVIDENT II study. Eur J Cardiovasc Nurs. 2018 Aug;17(6):552-562. doi: 10.1177/1474515118761870. Epub 2018 Feb 28. PMID 29488798
- [Derived] Recio-Rodriguez JI, Agudo-Conde C, Martin-Cantera C, Gonzalez-Viejo MN, Fernandez-Alonso MD, Arietaleanizbeaskoa MS, Schmolling-Guinovart Y, Maderuelo-Fernandez JA, Rodriguez-Sanchez E, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Investigators. Short-Term Effectiveness of a Mobile Phone App for Increasing Physical Activity and Adherence to the Mediterranean Diet in Primary Care: A Randomized Controlled Trial (EVIDENT II Study). J Med Internet Res. 2016 Dec 19;18(12):e331. doi: 10.2196/jmir.6814. PMID 27993759
- [Derived] Sanchez-Aguadero N, Alonso-Dominguez R, Recio-Rodriguez JI, Patino-Alonso MC, Gomez-Marcos MA, Martin-Cantera C, Schmolling-Guinovart Y, Garcia-Ortiz L; EVIDENT II Group. Dietary glycemic index and retinal microvasculature in adults: a cross-sectional study. Nutr J. 2016 Oct 18;15(1):88. doi: 10.1186/s12937-016-0209-2. PMID 27756385
- [Derived] Recio-Rodriguez JI, Martin-Cantera C, Gonzalez-Viejo N, Gomez-Arranz A, Arietaleanizbeascoa MS, Schmolling-Guinovart Y, Maderuelo-Fernandez JA, Perez-Arechaederra D, Rodriguez-Sanchez E, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Group. Effectiveness of a smartphone application for improving healthy lifestyles, a randomized clinical trial (EVIDENT II): study protocol. BMC Public Health. 2014 Mar 15;14:254. doi: 10.1186/1471-2458-14-254. PMID 24628961
- See also: Click here for more information about this study — https://apisal.es/